CLINICAL TRIAL: NCT07303751
Title: HPV Vaccination and Infectivity Reduction in HPV-positive Women
Brief Title: Study Assessing Reduced HPV Infectivity and Transmission in HPV-Positive Women Following Vaccination With 9vHPV
Acronym: RIFT-SSA
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Institut d'Investigació Biomèdica de Bellvitge (Other)
Responsible Party: Principal Investigator, Miquel Angel Pavon Ribas, Chief of Infection and Cancer Laboratory. Principal Investigator-PHD, Institut d'Investigació Biomèdica de Bellvitge
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: INV-074218
Record Dates: First submitted 2025-11-20; First posted 2025-12-26 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2026-02

CONDITIONS: HPV; High-risk HPV (Any Strain); Human Papillomavirus (HPV) Infections
Keywords: Cervical cancer; Cervical Intraepithelial Neoplasia Grade I/ II/ III (CIN I/II/III); Squamous Intraepithelial Lesions of the Cervix, High/ Low Grade; Human Papillomavirus (HPV) Infections; High-risk HPV; HPV-16/ 18; HPV DNA Tests; HPV Vaccines; HPV Nonavalent Vaccine; Gardasil-9; 9vHPV
MeSH Terms: conditions — Papillomavirus Infections; Infections; Uterine Cervical Neoplasms; Squamous Intraepithelial Lesions of the Cervix

STUDY DESIGN:
Intervention Model Description: This is randomized trial with two arms. First arm will receive one dose of the nonavalent vaccine and the second unvaccined arm will serve as a control.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervantional Arm (Experimental): Women randomisied on this arm will receive their first dose at Month 0 (M0).
  Interventions: Biological: Nonavalent HPV vaccine (9vHPV)
- Control Arm (No Intervention): Women randomised on this arm will not to be vaccinated at Month 0 (M0).

INTERVENTIONS:
Biological: Nonavalent HPV vaccine (9vHPV) — Nonavalent HPV vaccine (9vHPV/ Gardasil-9™). Sterile suspension, 0.5 ml dose, intramuscular, prepared from the highly purified viruslike particles (VLPs) of the major capsid L1 protein from 9 HPV types: 6/11/16/18/31/33/45/52/58. 9vHPV is currently indicated in the EU in individuals from 9 years of age for the prevention of diseases caused by vaccine's 9 HPV types: genital warts (HPV6 and 11) and premalignant lesions and cancers affecting the cervix, vulva, vagina and anus (HPV16, 18, 31, 22, 45, 52 and 58). It was authorized for marketing in the EU on June 9th, 201
  Other Names: Gardasil-9™
  Arms: Intervantional Arm

SUMMARY:
This is a randomized, open-label trial, to assess whether a single dose of HPV nonavalent vaccine, administered to HIV uninfected, unvaccinated women with high risk HPV16/18/31/33/45/52 or 58 can decrease the infectivity of shed HPV viruses.

Our hypothesis is that vaccination will have little or no impact on HPV sample positivity by DNA PCR since the viral particles will continue to be produced and released, but that particles will be neutralized by vaccine-induced antibodies, thereby reducing their infective capacity. Cervical samples will be collected at randomisation and at 6 months, to compare infectivity of shed HPV viruses.

ELIGIBILITY:
Inclusion Criteria:

* Born female
* Aged between 18-29 years old;
* Living in Kambia district (or neighbouring district if included) without plans to move away in the next 12 months;
* Willing to participate in the study and have signed the informed consent form;
* In good health as determined by a medical history (a physical examination will be conducted if necessary according to the clinician's judgement);
* Willing to be tested for HIV;
* Are HIV negative at the screening visit;
* Not pregnant;
* Able to pass a Test of Understanding (TOU);
* Willing to provide cervical, urine and blood samples;
* Agree to be vaccinated with a single dose of Gardasil9® if randomised to the vaccine arm at Day 0;
* Have no visible suspicious cervical lesions on examination.
* Agree to a pregnancy test at screening and before any HPV vaccination.

Exclusion Criteria:

* They have been previously vaccinated against HPV;
* They have a chronic condition, such as autoimmune conditions, degenerative diseases, neurologic or genetic diseases among others;
* They are HIV positive or immunocompromised;
* They are pregnant or planning to get pregnant in the next 12 months;
* They are less than three months post-partum or currently breastfeeding;
* They are allergic to one of the vaccine components or to latex;
* They are sexually active and are not using, or are not willing to use, an effective birth control method from D-14 until 60 days after the last vaccine dose
* The nurse or clinician determining the eligibility, in agreement with principal investigator, considers that there is a reason that precludes participation.

Ages: 18 Years to 29 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — We will enroll only ciswomen
Enrollment: 80 (Estimated)
Dates: Start 2026-02-01 (Estimated); Primary Completion 2027-02-01 (Estimated); Study Completion 2027-02-01 (Estimated)

PRIMARY OUTCOMES:
The difference in infective capacity of cervical HPV virions at 6 months, between HPV-positive unvaccinated women and HPV-positive women who receive one dose of the HPV L1 nonavalent vaccine (Gardasil9®). | 7 months
  To analyse the differences in the HPV neutralization capacity of HPV 16, 18, 31, 33, 45, 52, 58 vaccine-induced antibodies in serum and cervical samples at month 6 between HPV-positive unvaccinated women and HPV-positive women who receive one dose of the HPV L1 nonavalent vaccine (Gardasil9®).

SECONDARY OUTCOMES:
The difference in the HPV neutralization capacity of vaccine-induced antibodies in serum and cervical samples at 6 months, between HPV-positive unvaccinated women with HPV-positive women who receive one dose of the HPV L1 nonavalent vaccine | 7 months
  To analyse the differences in the HPV neutralization capacity of HPV 16, 18, 31, 33, 45, 52, 58 vaccine-induced antibodies in serum and cervical samples at month 6 between HPV-positive unvaccinated women and HPV-positive women who receive one dose of the HPV L1 nonavalent vaccine (Gardasil9®).
The difference in HPV viral load in cervical samples at 6 months, between HPV-positive unvaccinated women with HPV-positive women who receive one dose of the HPV L1 nonavalent vaccine (Gardasil9®). | 7 months
  To analyse the differences in the HPV viral load in cervical samples at 6 months between HPV-positive unvaccinated women and HPV-positive women who receive one dose of the HPV L1 nonavalent vaccine (Gardasil9®).
Neutralising antibodies infective capacity of HPV virions and HPV viral load in urine samples | 7 months
  To analyse urine samples at month 6 to detect neutralizing antibodies to HPV 16, 18, 31, 33, 45, 52, 58, and the infective capacity of HPV 16, 18, 31, 33, 45, 52, 58 virions and to measure HPV 16, 18, 31, 33, 45, 52, 58 viral load
The difference in infectivity reduction and vaccine induced antibodies among different HPV types. | 7 months
  To analyse differences in infectivity reduction and vaccine induced antibodies among different HPV types included in the 9-valent vaccine.

CONTACTS AND LOCATIONS:
Locations (1):
- Kambia Research Centre, Freetown, Sierra Leone

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hooper R, Forbes A, Hemming K, Takeda A, Beresford L. Analysis of cluster randomised trials with an assessment of outcome at baseline. BMJ. 2018 Mar 20;360:k1121. doi: 10.1136/bmj.k1121. No abstract available. PMID 29559436
- [Background] Houlihan CF, Baisley K, Bravo IG, Kapiga S, de Sanjose S, Changalucha J, Ross DA, Hayes RJ, Watson-Jones D. Rapid acquisition of HPV around the time of sexual debut in adolescent girls in Tanzania. Int J Epidemiol. 2016 Jun;45(3):762-73. doi: 10.1093/ije/dyv367. Epub 2016 Mar 4. PMID 26944311
- [Background] Centers for Disease Control and Prevention. (2025, 6 de marzo). Human Papillomavirus (HPV) Vaccine Safety. https://www.cdc.gov/vaccine-safety/vaccines/hpv.html
- [Background] Watson-Jones D, Baisley K, Brown J, Kavishe B, Andreasen A, Changalucha J, Mayaud P, Kapiga S, Gumodoka B, Hayes RJ, de Sanjose S. High prevalence and incidence of human papillomavirus in a cohort of healthy young African female subjects. Sex Transm Infect. 2013 Aug;89(5):358-65. doi: 10.1136/sextrans-2012-050685. Epub 2013 Mar 13. PMID 23486859
- [Background] Centers for Disease Control and Prevention. (2024, 9 de julio). HPV Vaccine Safety and Effectiveness Data. https://www.cdc.gov/hpv/hcp/vaccination-considerations/safety-and-effectiveness-data.html
- [Background] Chow EP, Read TR, Wigan R, Donovan B, Chen MY, Bradshaw CS, Fairley CK. Ongoing decline in genital warts among young heterosexuals 7 years after the Australian human papillomavirus (HPV) vaccination programme. Sex Transm Infect. 2015 May;91(3):214-9. doi: 10.1136/sextrans-2014-051813. Epub 2014 Oct 10. PMID 25305210
- [Background] Whitworth HS, Mounier-Jack S, Choi EM, Gallagher KE, Howard N, Kelly H, Mbwanji G, Kreimer AR, Basu P, Barnabas R, Drolet M, Brisson M, Watson-Jones D. Efficacy and immunogenicity of a single dose of human papillomavirus vaccine compared to multidose vaccination regimens or no vaccination: An updated systematic review of evidence from clinical trials. Vaccine X. 2024 Apr 16;19:100486. doi: 10.1016/j.jvacx.2024.100486. eCollection 2024 Aug. PMID 38873638
- [Background] Kamolratanakul S, Pitisuttithum P. Human Papillomavirus Vaccine Efficacy and Effectiveness against Cancer. Vaccines (Basel). 2021 Nov 30;9(12):1413. doi: 10.3390/vaccines9121413. PMID 34960159
- [Background] Sung H, Ferlay J, Siegel RL, Laversanne M, Soerjomataram I, Jemal A, Bray F. Global Cancer Statistics 2020: GLOBOCAN Estimates of Incidence and Mortality Worldwide for 36 Cancers in 185 Countries. CA Cancer J Clin. 2021 May;71(3):209-249. doi: 10.3322/caac.21660. Epub 2021 Feb 4. PMID 33538338
- [Background] Teblick L, Lipovac M, Molenberghs F, Delputte P, De Vos WH, Vorsters A. HPV-specific antibodies in female genital tract secretions captured via first-void urine retain their neutralizing capacity. Hum Vaccin Immunother. 2024 Dec 31;20(1):2330168. doi: 10.1080/21645515.2024.2330168. Epub 2024 Apr 3. PMID 38567541
- [Background] Smahelova J, Hamsikova E, Ludvikova V, Vydrova J, Traboulsi J, Vencalek O, Lukes P, Tachezy R. Outcomes After Human Papillomavirus Vaccination in Patients With Recurrent Respiratory Papillomatosis: A Nonrandomized Clinical Trial. JAMA Otolaryngol Head Neck Surg. 2022 Jul 1;148(7):654-661. doi: 10.1001/jamaoto.2022.1190. PMID 35653138
- [Background] Wenande E, Hastrup A, Wiegell S, Philipsen PA, Thomsen NB, Demehri S, Kjaer SK, Haedersdal M. Human Papillomavirus Vaccination and Actinic Keratosis Burden: The VAXAK Randomized Clinical Trial. JAMA Dermatol. 2025 Jun 1;161(6):605-614. doi: 10.1001/jamadermatol.2025.0531. PMID 40047786
- [Background] Drolet M, Benard E, Perez N, Brisson M; HPV Vaccination Impact Study Group. Population-level impact and herd effects following the introduction of human papillomavirus vaccination programmes: updated systematic review and meta-analysis. Lancet. 2019 Aug 10;394(10197):497-509. doi: 10.1016/S0140-6736(19)30298-3. Epub 2019 Jun 26. PMID 31255301